CLINICAL TRIAL: NCT05748054
Title: Early Childhood Caries in Jordanian Children: Prevalence, Risk Factors and Prevention Using Silver Diamine Fluoride
Brief Title: Early Childhood Caries in Jordanian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 47/2019
Record Dates: First submitted 2023-02-05; First posted 2023-02-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Early Childhood Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Children who receive a single application of 38% SDF
  Interventions: Drug: Silver Diamine Fluoride
- Control group (No Intervention): Children do not receive any intervention

INTERVENTIONS:
Drug: Silver Diamine Fluoride — A colourless solution known with its alkaline nature; it simply consists of a union of silver, fluoride and ammonia. It can be applied on caries cavities using a micro-brush.
  Other Names: SDF
  Arms: Study group

SUMMARY:
In this cross sectional epidemiological study, we aimed to report the prevalence of early childhood caries (ECC) in children attending kindergartens in Jordan, and its associated risk factors. We also, aimed to determine the effectiveness of silver diamine fluoride as a caries control material and its acceptance among parents of children with ECC. Children (n=887) with mean age 4.64 ± 1.56 were examined. Among this sample there was a number of children (n=159) who were enrolled in a randomized controlled trial to study silver diamine fluoride efficacy in caries control. The sample consisted of two groups; the study group (children who received single spot application of 38% SDF) and control group (children who were examined only).

DETAILED DESCRIPTION:
Background: Early childhood caries is a well-known international public health challenge amongst young children.

Aims: To report the prevalence of early childhood caries in children attending kindergartens in Jordan, and its associated risk factors. To determine the effectiveness of silver diamine fluoride as a caries control material and its acceptance among parents of children with ECC.

Methods: This is a cross sectional epidemiological study comprised of children (n=887) with mean age 4.64 ± 1.56 who attended kindergartens of different cities in Jordan, this sample received questionnaires to fill data related to their demographic, socioeconomic, oral hygiene, oral health, nursing and nutritional habits. These children were also examined to determine early childhood caries prevalence in Jordan. Among this sample there was a number of children (n=159) with the mean age 4.8 ± 0.85 who were planned to be involved in a sample of a randomized controlled trial to study silver diamine fluoride efficacy in caries control. The sample consisted of two groups; the study group (children who received single spot application of 38% SDF) and control group (children who were examined only). Application of SDF started after distribution and receiving back approval letters from children's parents accompanied with questionnaires for data related to the approval/disapproval of the application. The sample were followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Children with early childhood caries involving anterior and/or posterior primary teeth
* Children with with cavitated lesions with active caries
* Children with no clinical signs of pulp involvement

Exclusion criteria:

* Children with grossly broken down teeth
* Children with teeth with more than one third of the crown missing
* Children with pulpally involved teeth (with pulp exposure, presence of an abscess or a sinus) Children with obvious discoloration, and abnormal mobility

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of early childhood caries | After 1 year
  The percentage of children with early childhood caries
Caries Prevention | After 1 year of SDF application
  Prevention of new cavities
Caries arrest | After 1 year of SDF application
  Arrest of existing cavities

SECONDARY OUTCOMES:
Risk factors for early childhood caries | After 1 year
  Early childhood caries risk factors questionnaire
Parental acceptance of SDF | Before application of SDF
  Reasons for acceptance or unacceptance of SDF application

CONTACTS AND LOCATIONS:
Overall Officials: Ola B. Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llodra JC, Rodriguez A, Ferrer B, Menardia V, Ramos T, Morato M. Efficacy of silver diamine fluoride for caries reduction in primary teeth and first permanent molars of schoolchildren: 36-month clinical trial. J Dent Res. 2005 Aug;84(8):721-4. doi: 10.1177/154405910508400807. PMID 16040729
- [Background] Mei ML, Chu CH, Low KH, Che CM, Lo EC. Caries arresting effect of silver diamine fluoride on dentine carious lesion with S. mutans and L. acidophilus dual-species cariogenic biofilm. Med Oral Patol Oral Cir Bucal. 2013 Nov 1;18(6):e824-31. doi: 10.4317/medoral.18831. PMID 23722131
- [Background] Ramos-Gomez FJ, Shepard DS. Cost-effectiveness model for prevention of early childhood caries. J Calif Dent Assoc. 1999 Jul;27(7):539-44. PMID 10530112
- [Background] Zhi QH, Lo EC, Lin HC. Randomized clinical trial on effectiveness of silver diamine fluoride and glass ionomer in arresting dentine caries in preschool children. J Dent. 2012 Nov;40(11):962-7. doi: 10.1016/j.jdent.2012.08.002. Epub 2012 Aug 11. PMID 22892463
- [Background] Gao SS, Zhang S, Mei ML, Lo EC, Chu CH. Caries remineralisation and arresting effect in children by professionally applied fluoride treatment - a systematic review. BMC Oral Health. 2016 Feb 1;16:12. doi: 10.1186/s12903-016-0171-6. PMID 26831727